CLINICAL TRIAL: NCT04217070
Title: Evaluation of Suicidal Poisoning Cases in Emergency Units of Assuit University Hospitals
Brief Title: Suicidal Poisoning in Emergency Units
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Gehad Hussien Eisa, principle investigator, Assiut University
Other Study IDs: ESPEUAUH
Record Dates: First submitted 2019-12-31; First posted 2020-01-03 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Poisoning
MeSH Terms: conditions — Poisoning | interventions — Surveys and Questionnaires; Blood Gas Analysis; epicatechin gallate; Mass Screening

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Questionnaire including demographic data, data regarding poisoning substance and outcomes of suicidal attempts
  Other Names: ABG, ECG, ECHO, SCREENING TESTS

SUMMARY:
Poisoning is the deterioration of the body's functions by the ingestion of any substance being toxic to the body or by overdosing a nontoxic substance. Poisoning cases may vary according to the geographical and seasonal characteristics of the region, sociocultural structure of the population, life index and the age groups.

Worldwide, intentional self-poisoning (ISP) is the most common form of suicide attempt and the most common method that results in medical hospitalization.

DETAILED DESCRIPTION:
Questionnaire is prepared including the following items:

Demographic data:

Gender -age-marital status -occupation- socioeconomic state -special habit -history of psychiatric innless-history of chronic diseases-history of drug dependence -previous suicidal attempts-toxic substance used in suicide- time of poisoning, season and time of arrival .

Data regarding poisoned substance:

Dose, type of the substance used and rout of administration. Presenting symptoms of intoxication and management

Complete clinical examination:

General condition: conscious level and vital signs. Local examination: chest, heart, abdomen, etc.

Investigation:

(Arterial blood gases - ECG -otherwise according to case presentation)

Prognosis:

Complete recovery, complications, death.

ELIGIBILITY:
Inclusion Criteria:

* suicidal poisoning cases

Exclusion Criteria:

* other causes of suicide

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All patients presented to Emergency units of assiut university hospitals with suicidal poisoning attemps
Sampling Method: Probability Sample
Enrollment: 303 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Determination of the prevalence of suicidal poisoning cases attending emergency units, Assuit university hospitals | One year
  Number of cases of all age group committing suicide by poisoning in a peroid of one year will be known. accidental poisoning will be detected to release the prevalence of suicidal poisoning

CONTACTS AND LOCATIONS:
Overall Officials: Randa H Abd-Elhady, prof, Study Director; Noha E Ebrahem, Dr, Study Director
Locations (1):
- Assiut University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Conner KR, Wiegand TJ, Gorodetsky R, Schult RF, Kaukeinen K. Poisoning Severity Associated with a Range of Medications in Suicide Attempts by Ingestion. Suicide Life Threat Behav. 2019 Jun;49(3):635-642. doi: 10.1111/sltb.12468. Epub 2018 Apr 25. PMID 29693268
- [Background] Kanchan T, Menezes RG. Suicidal poisoning in Southern India: gender differences. J Forensic Leg Med. 2008 Jan;15(1):7-14. doi: 10.1016/j.jflm.2007.05.006. Epub 2007 Sep 5. PMID 18096509
- [Background] Kazanasmaz H, Kazanasmaz O, Calik M. Epidemiological and sociocultural assessment of childhood poisonings. Turk J Emerg Med. 2019 Jun 20;19(4):127-131. doi: 10.1016/j.tjem.2019.06.001. eCollection 2019 Oct. PMID 31687610
- [Background] Piekarska-Wijatkowska A, Kobza-Sindlewska K, Rogaczewska A, Zajdel R, Krakowiak A. Intentional poisoning among elderly people-residents of a large urban agglomeration in Poland. Hum Exp Toxicol. 2016 Dec;35(12):1328-1336. doi: 10.1177/0960327116630353. Epub 2016 Feb 9. PMID 26860687
- [Background] Klonsky ED, May AM, Saffer BY. Suicide, Suicide Attempts, and Suicidal Ideation. Annu Rev Clin Psychol. 2016;12:307-30. doi: 10.1146/annurev-clinpsy-021815-093204. Epub 2016 Jan 11. PMID 26772209